CLINICAL TRIAL: NCT07073040
Title: Efficacy and Safety of Cold Atmospheric Plasma Combined With Endovascular Intervention in Patients With Diabetic Foot Ulcers and Lower Extremity Arterial Occlusion: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Cold Atmospheric Plasma Combined With Endovascular Intervention in Patients With Diabetic Foot Ulcers and Lower Extremity Arterial Occlusion
Acronym: PROSPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: Ansteel General Hospital (Unknown); Tsinghua University (Other)
Responsible Party: Principal Investigator, Lin Tao, Associate Professor, Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROSPECT
Record Dates: First submitted 2025-06-29; First posted 2025-07-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcers (DFU); Lower Extremity Arterial Occlusion
Keywords: cold atmospheric plasma; diabetic foot ulcers; lower extremity arterial occlusion
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants in the placebo group will undergo a sham procedure, in which the electric field required for plasma generation will be disabled, so that no plasma is produced. Only the operating sounds of the device will be simulated, ensuring blinding for both participants and clinical staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAP therapy (Active Comparator)
  Interventions: Device: Cold atmospheric plasma (CAP); Other: Successful infrapopliteal angioplasty
- the placebo group (Placebo Comparator)
  Interventions: Device: Sham Procedure; Other: Successful infrapopliteal angioplasty

INTERVENTIONS:
Device: Cold atmospheric plasma (CAP) — CAP therapy will be administered once daily for the first five days and then every other day thereafter, for a total of 13 sessions. Each session will last approximately 25 minutes, as recommended by the manufacturer. During treatment, the affected limb will be enclosed in a sterile treatment bag, sealed with medical adhesive tape. The CAP device will operate in two sequential modes: a "disinfection mode" delivering ozone-rich (O₃) plasma-activated gas for 20 minutes, followed by a "healing mode" delivering nitric oxide (NO)-rich plasma-activated gas for 5 minutes. All procedures will be performed in accordance with the manufacturer's instructions and the device's standard operating protocol.
  Arms: CAP therapy
Device: Sham Procedure — Participants in the placebo group will undergo a sham procedure, in which the electric field required for plasma generation will be disabled, so that no plasma will be produced. Only the operating sounds of the device will be simulated, ensuring blinding for both participants and clinical staff.
  Arms: the placebo group
Other: Successful infrapopliteal angioplasty — All patients will undergo successful infrapopliteal angioplasty, with less than 30% residual stenosis confirmed by digital subtraction angiography.

SUMMARY:
Critical limb ischemia is the end-stage manifestation of peripheral arterial disease (PAD), frequently presenting as ischemic rest pain, ulceration, or gangrene. Diabetes mellitus is a major risk factor for lower extremity arterial occlusion, with infrapopliteal arteries most commonly affected. Patients with diabetic foot ulcers (DFUs) have a high prevalence of neurovascular complications, poor healing, and elevated amputation and mortality rates. Large-scale cohort studies indicate that five-year survival after amputation in this population is only about 50%, underscoring the need for more effective therapies.

Endovascular revascularization has become the first-line treatment for diabetic lower limb ischemia. However, despite successful revascularization, persistent microvascular dysfunction and difficult-to-heal ulcers remain common due to chronic inflammation, impaired angiogenesis, and tissue repair deficits. Current advanced wound dressings provide limited benefit and are often costly.

Cold atmospheric plasma (CAP) has emerged as a promising adjunctive therapy, with demonstrated antimicrobial activity-including efficacy against multidrug-resistant organisms-and the ability to promote microcirculation and wound healing. CAP generates reactive oxygen and nitrogen species that disrupt bacterial membranes and may also stimulate tissue regeneration. Preclinical and clinical studies suggest that CAP can accelerate healing in chronic wounds and is well tolerated by patients.

Given these advantages, the present study aims to assess the efficacy and safety of CAP combined with endovascular intervention in patients with diabetic foot ulcers and lower extremity arterial occlusion, to inform future clinical application of this novel technology.

DETAILED DESCRIPTION:
End-stage peripheral arterial disease (PAD) is characterized by critical limb ischemia, which manifests clinically as insufficient arterial perfusion leading to ischemic rest pain, ulceration, and gangrene. A substantial proportion of these cases occur in patients with diabetes complicated by lower extremity arterial occlusion. Ischemia in diabetic patients predominantly affects infrapopliteal arteries, often presenting bilaterally and symmetrically, with diffuse lesions that commonly involve the entire vessel wall. These patients are more prone to both intimal atherosclerosis and medial arterial calcification.

A large multicenter cohort study in China that enrolled 669 patients with diabetic foot ulcers from 15 tertiary hospitals reported that more than 98% had underlying neurovascular pathology. The overall amputation rate was 19.03%, with major and minor amputation rates of 2.14% and 16.88%, respectively. Notably, the five-year survival rate after amputation was approximately 50%, which is lower than that observed for many malignancies. According to a large European cohort study, about half of diabetic foot ulcers are attributable to neuropathic or ischemic etiologies. Both macrovascular and microvascular dysfunctions jointly impair tissue perfusion and exacerbate diabetic foot pathology. From a clinical perspective, successful arterial revascularization alone is not sufficient; maintenance and optimization of distal microcirculatory perfusion following revascularization are also essential for effective ulcer healing.

With advances in endovascular techniques, infrapopliteal angioplasty has become the first-line treatment for diabetic lower limb ischemia, with proven efficacy. However, even after successful revascularization, some patients continue to suffer from inadequate distal perfusion due to microembolization or from persistent, hard-to-heal ulcers driven by the underlying pathophysiology of diabetic wounds. Several studies have demonstrated that diabetic patients experience metabolic dysregulation, local wound hyperglycemia, and accumulation of advanced glycation end-products (AGEs); combined with immune dysfunction and chronic inflammation, these factors maintain wounds in a persistent inflammatory state. Chronic inflammation suppresses vascular endothelial growth factor (VEGF) and angiopoietin-1 (ANG-1) expression, impairs endothelial cell function, and leads to angiogenesis disorders and delayed tissue repair. Reduced VEGF and ANG-1 expression has been confirmed in skin specimens from diabetic patients. In addition, peripheral neuropathy further inhibits neovascularization.

Despite widespread clinical use of advanced wound dressings-such as hydrogels, natural or synthetic polymer-based products, and other dressings designed specifically for diabetic ulcers-treatment efficacy remains limited, and costs can be substantial. For patients with diabetic foot ulcers complicated by large-vessel occlusion, ongoing assessment and support of distal microvascular perfusion remain a major unmet clinical need, even after successful revascularization.

Cold atmospheric plasma (CAP) has been widely adopted in medical applications and has demonstrated robust antimicrobial activity as well as the capacity to enhance tissue microcirculation and promote wound healing, with excellent patient tolerance. Multiple preclinical and clinical studies have confirmed the bactericidal efficacy of CAP, including activity against multidrug-resistant organisms. For example, Brun et al. reported that CAP effectively eradicates Pseudomonas aeruginosa and methicillin-resistant Staphylococcus aureus (MRSA) in vitro, achieving results comparable to antibiotics but with higher efficiency. Lis et al. found that CAP could also inactivate MRSA, Klebsiella pneumoniae, and Acinetobacter baumannii. Korean researchers Kim et al. demonstrated that CAP effectively disrupts biofilms formed by P. aeruginosa and other pathogens in canine skin and ear infections. In a prospective clinical study, Stratmann et al. showed that CAP treatment accelerates wound healing in diabetic foot ulcers. Boekema et al. [6] reported a significant reduction in bacterial load and no serious adverse events in patients with P. aeruginosa infections treated with CAP, confirming its safety profile.

The antimicrobial mechanism of CAP is primarily attributed to the generation of reactive oxygen and nitrogen species (RONS), which induce local free radical formation and disrupt microbial membranes, leading to apoptosis without fostering antimicrobial resistance. This highlights CAP as a valuable adjunct to conventional antibiotic therapy, especially for wounds infected with multidrug-resistant bacteria.

Importantly, CAP's benefits extend beyond antimicrobial effects. Numerous studies indicate that CAP promotes wound healing not only by eliminating pathogens but also by directly activating tissue regeneration. At the cellular level, CAP has been shown to modulate fibroblasts, vascular endothelial cells, and keratinocytes. Stratmann et al. observed that CAP enhanced tissue regeneration in diabetic foot ulcers without a corresponding decrease in colony-forming units, suggesting a regeneration mechanism independent of bactericidal action. In the study by Brehmer et al., CAP (PlasmaDerm device) significantly improved healing rates in lower extremity venous ulcers compared with standard care. These findings imply that CAP can accelerate tissue regeneration and shorten healing time, regardless of its antimicrobial effects.

Delayed wound healing is often accompanied by local microcirculatory disorders, resulting in decreased collagen production and impaired proliferation and migration of keratinocytes and fibroblasts. Several clinical trials have demonstrated that CAP exposure at therapeutic doses increases local skin blood flow and tissue oxygen saturation without raising skin temperature. The underlying mechanism may involve nitric oxide (NO) permeation, modulation of cysteine disulfide bonds and acidic lipid groups, reduced local pH, and improved microcirculation. In animal and cellular experiments, Arndt et al. demonstrated that CAP induces oxidative stress pathways in a paracrine and autocrine manner, stimulating keratinocytes, fibroblasts, and endothelial cells to produce vascular growth factors (EGF, FGF-2, IL-8, uPA, angiopoietin, VEGF), thereby promoting angiogenesis.

Based on these findings, this study aims to evaluate the efficacy and safety of CAP combined with endovascular intervention in patients with diabetic foot ulcers complicated by lower extremity arterial occlusion, providing essential evidence to support future large-scale clinical application of CAP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years, with a diagnosis of type 1 or type 2 diabetes and diabetic foot ulcer; glycated hemoglobin (HbA1c) ≤ 10%.
* Presence of at least one chronic foot ulcer persisting for at least three weeks, with no signs of healing after standard-of-care treatment based on current clinical guidelines. The ulcer must be classified as Wagner-Armstrong grade 1D or 2D (Wagner: superficial ulcer [grade 1] or ulcer extending to tendon [grade 2]; Armstrong: presence of both ischaemia and infection [stage D]).
* Documented infrapopliteal arterial stenosis or occlusion by vascular ultrasound and/or CT angiography (CTA), meeting indications for revascularization. All enrolled patients must have received successful infrapopliteal balloon angioplasty, with intraoperative angiography confirming target artery patency.
* Provision of written informed consent.

Exclusion Criteria:

* Concurrent treatment of the wound with local vacuum therapy or maggot therapy.
* Undergoing dialysis.
* Use of local active antibiotics.
* Treatment with platelet-rich fibrin.
* Women of childbearing potential without effective contraception, or women who are actively breastfeeding.
* Presence of other severe organ dysfunction, with an expected survival of less than six months.
* Participation in another clinical trial within the past three months or currently enrolled in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
Change in ulcer area between groups | From Baseline (Day 0) to Day 21 post-randomization
  The ulcer area (cm²) will be measured daily during the first five days, and every other day for the subsequent eight visits (13 follow-up assessments in total)

SECONDARY OUTCOMES:
Time to 10% reduction in ulcer area | From Baseline (Day 0) to Day 21 post-randomization
  The time from randomization to the first occurrence of a 10% reduction in ulcer area
Time to 20% reduction in ulcer area | From Baseline (Day 0) to Day 21 post-randomization
  The time from randomization to the first occurrence of a 20% reduction in ulcer area.
Time to onset of clinical signs of infection | From Baseline (Day 0) to Day 21 post-randomization
  The time from randomization to the first documented clinical sign of wound infection.
Change in pain score | From Baseline (Day 0) to Day 21 post-randomization
  Change in pain score, assessed by the Visual Analogue Scale (VAS; 0 = no pain, 10 = worst imaginable pain; higher scores indicate greater pain severity)
Change in quality of life (EQ-5D questionnaire) | Baseline (Day 0) and Day 21 post-randomization
Change in quality of life (SF-12 questionnaire) | Baseline (Day 0) and Day 21 post-randomization
Incidence of local skin irritation | From Baseline (Day 0) to Day 21 post-randomization
Incidence of local bleeding | From Baseline (Day 0) to Day 21 post-randomization
Incidence of local burning sensation | From Baseline (Day 0) to Day 21 post-randomization

OTHER OUTCOMES:
Change in pain score | Baseline (Day 0), Day 180 ± 15, and Day 360 ± 20 post-randomization
Change in quality of life (EQ-5D questionnaire) | Baseline (Day 0), Day 180 ± 15, and Day 360 ± 20 post-randomization
Change in quality of life (SF-12 questionnaire) | Baseline (Day 0), Day 180 ± 15, and Day 360 ± 20 post-randomization
Incidence of keloid formation | Baseline (Day 0), Day 180 ± 15, and Day 360 ± 20 post-randomization
Incidence of amputation | Baseline (Day 0), Day 180 ± 15, and Day 360 ± 20 post-randomization
All-cause mortality | Baseline (Day 0), Day 180 ± 15, and Day 360 ± 20 post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Yun-En Liu, MD, Study Chair — Shenyang Medical College; Lin Tao, MM, Principal Investigator — Shenyang Medical College
Locations (1):
- Ansteel General Hospital, Anshan, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol